CLINICAL TRIAL: NCT06967103
Title: QL1706 Combined With PE Compared With PE for the Neoadjuvant Treatment of HR+/HER2- Breast Cancer
Brief Title: QL1706 for the Neoadjuvant Treatment of HR+/HER2- Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-024
Record Dates: First submitted 2025-04-30; First posted 2025-05-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; HR+/HER2- Breast Cancer
Keywords: PD1; CTLA4; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 group (Experimental): NabPE+QL1706 every 3 weeks for 6 cycles. Then participants will receive surgery and QL1706 will be given as monotherapy every 3 weeks up to 6 months from the beginning of the treatment.
  Interventions: Drug: QL1706; Drug: Nab-PE
- NabPE group (Active Comparator): NabPEevery 3 weeks for 6 cycles. Then participants will receive surgery

INTERVENTIONS:
Drug: QL1706 — bispecific antibody targeting PD-1 and CLTA-4
  Arms: QL1706 group
Drug: Nab-PE — Nab-paclitaxel+Epirubicin
  Arms: QL1706 group

SUMMARY:
The goal of this clinical trial is to learn if QL1706 is effective in early HR+/HER2- breast cancer. It will also learn about the safety of QL1706. The main questions it aims to answer are:

Does QL1706 combined with neoadjuvant chemotherapy improve the pCR rate of early HR+/HER2- breast cancer? What adverse events do participants have when receiving QL1706? Participants will: Receive QL1706 plus chemotherapy or chemotherapy every 3 weeks for 6 cycles; All patients will receive surgery, and the primary end point is pathological complete response at the time of definitive surgery; After definitive surgery, the participants will receive adjuvant QL1706 every 3 weeks for up to 6 months from the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria

Subjects meeting all of the following criteria are eligible for inclusion in this study:

Voluntarily participates in the study, signs the informed consent form, and demonstrates good compliance.

Female, aged ≥18 years .

Evaluated by the research center as eligible to tolerate and scheduled to undergo radical breast cancer surgery, with no prior systemic anti-tumor therapy for breast cancer.

cT2 - T4d N0-N3, or cT1c with axillary lymph node metastasis confirmed clinically and pathologically；

Histologically and/or cytologically confirmed hormone receptor-positive (HR+) breast cancer (estrogen receptor [ER] or progesterone receptor [PR] nuclear staining >1%) with Ki67 ≥20%.

HER2-negative breast cancer, defined as:

Negative in situ hybridization (ISH) results; or

Immunohistochemistry (IHC) status of 0, 1+, or 2+. If IHC is 2+, ISH (e.g., FISH, CISH, SISH) must be negative.

Willing to provide fresh or archived tumor tissue samples.

At least one measurable lesion per RECIST 1.1 criteria.

Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Adequate organ function, defined as:

Hematology:

Hemoglobin ≥90 g/L

Absolute neutrophil count ≥1.5 × 10⁹/L

Platelet count ≥100 × 10⁹/L.

Biochemistry:

ALT and AST ≤2.5 × ULN (≤5 × ULN if liver metastases present);

Total bilirubin ≤1.5 × ULN;

Serum creatinine ≤1.5 × ULN or creatinine clearance (CCr) ≥60 mL/min.

Coagulation:

Activated partial thromboplastin time (APTT) ≤1.5 × ULN;

International normalized ratio (INR) ≤1.5 × ULN.

Cardiac function:

Left ventricular ejection fraction (LVEF) ≥50% by echocardiography.

Premenopausal or perimenopausal subjects must agree to use reliable and effective contraception or practice abstinence from the time of informed consent until at least 90 days after the last dose of study treatment.

Exclusion Criteria

Subjects meeting any of the following criteria will be excluded from this study:

Known severe hypersensitivity to macromolecular protein preparations, QL1706, albumin-bound paclitaxel, epirubicin hydrochloride, or their excipients.

Stage IV metastatic breast cancer or other conditions deemed ineligible for curative surgery after neoadjuvant therapy by the investigator.

Inflammatory breast cancer or bilateral primary breast cancer (including invasive or in situ carcinoma).

Major surgery or significant trauma within 28 days prior to the first dose.

Administration of live attenuated vaccines within 28 days before the first dose or anticipated during the study.

Systemic corticosteroids or immunosuppressive therapy within 14 days prior to the first dose or anticipated during the study.

Active autoimmune disease requiring systemic treatment within 2 years prior to enrollment, or history of autoimmune disorders.

Severe systemic infection within 28 days or active infection requiring intravenous/oral antibiotics within 14 days prior to the first dose.

Prior organ or allogeneic bone marrow transplantation or awaiting transplantation.

History or evidence of interstitial lung disease or active non-infectious pneumonitis.

Bleeding tendency or high risk of hemorrhage.

Thromboembolic events (e.g., cerebrovascular accident, pulmonary embolism) within 6 months prior to enrollment.

Congenital or acquired immunodeficiency (e.g., HIV infection).

Active hepatitis:

Hepatitis B: HBsAg-positive with HBV DNA ≥2000 IU/mL;

Hepatitis C: HCV antibody-positive with HCV RNA above the upper limit of normal.

Poorly controlled cardiac conditions, including:

NYHA Class II or higher heart failure or LVEF <50%;

Unstable angina;

Myocardial infarction within 1 year;

QTc interval >470 ms (female) on resting ECG.

Other malignancies within 5 years (excluding basal cell carcinoma or cervical carcinoma in situ).

Use of investigational drugs within 4 weeks prior to the first dose.

History or current diagnosis of neurological or psychiatric disorders (e.g., epilepsy, dementia).

History of pancreatitis.

Pregnancy, lactation, or refusal to use contraception.

Any other condition deemed inappropriate for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response | up to 24 weeks
  After neoadjuvant chemotherapy and surgery, the resected specimen (breast + axilla) was free of any invasive cancer (ie, ypT0/is, ypN0)
pathological complete response in PDL1 positive subgroup | up to 24 weeks
  After neoadjuvant chemotherapy and surgery, the resected specimen (breast + axilla) was free of any invasive cancer (ie, ypT0/is, ypN0)

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | 5-10 years
  Disease-free Survival,From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause
Objective Response Rate (ORR) | up to 24 weeks
  ORR is defined as proportion of patients demonstrating either a partial response (PR) or a complete response (CR)
adverse events | up to 24 weeks
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, China